CLINICAL TRIAL: NCT02100566
Title: Behavioral Economics for Advance Care OptioNs
Acronym: BEACON
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ascension Health (Industry)
Collaborators: University of Pennsylvania (Other); Robert Wood Johnson Foundation (Other)
Responsible Party: Principal Investigator, Mark Vogel, PhD, Director of Behavioral Science and Psychology, Ascension Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: RWJ 71476
Record Dates: First submitted 2014-03-27; First posted 2014-04-01 (Estimated); Last update posted 2021-07-27 (Actual); Status verified 2021-07

CONDITIONS: End of Life Care
Keywords: Advance Directive
MeSH Terms: interventions — Counseling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Behavioral Counseling (Experimental): Provide an advance directive document to patients along with counseling that either focuses on care giver burden or on patient autonomy.
  Interventions: Behavioral: Counseling (Care giver burden focus); Behavioral: Counseling (patient autonomy focus)
- Standard AD (No Intervention): The topic of advance directives (AD) is introduced but patient receives an AD document only upon request.

INTERVENTIONS:
Behavioral: Counseling (Care giver burden focus) — An advance directive (AD) document is provided to the patient along with counseling that focuses on care giver burden as the reason for adoption of the AD.
  Other Names: Focusing effect
  Arms: Behavioral Counseling
Behavioral: Counseling (patient autonomy focus) — An advance directive (AD) document is provided to the patient along with counseling that focuses on patient autonomy (control) as the reason for adoption of the AD.
  Other Names: Focusing effect
  Arms: Behavioral Counseling

SUMMARY:
People with life-limiting illness often receive more aggressive healthcare than desired including costly procedures that provide little medical benefit. Advance Directives (AD) can reduce this effect but various factors limit their adoption.

A randomized trial will target hospitalized patients with a serious, life limiting illness to test if the behavioral economics principles of endowment (possessing something) and focusing (featuring something important to patients) can motivate AD completion. Investigators will examine if offering patients an AD by default, in combination with framing the rationale for AD completion (emphasizing patient control or caregiver burden) improves AD completion and family conversation compared to a no-intervention group. The study hypothesis is to determine if rates of AD completion and family conversations will be highest among patients receiving the intervention focused on reduced caregiver burden; and if the two intervention groups will have higher rates of both than the control group.

The investigators suspect that a small change in how patient information is framed (endowment and focusing used in tandem) will potentially leverage large increases in AD completion and that targeting HHC patients allows AD discussions early in the disease trajectory when they can participate in care decisions.

DETAILED DESCRIPTION:
Primary research question: Does offering patients an Advance Directive (AD) document (by default), in combination with framing the rationale for AD completion (emphasizing either: A. patient control; or B. reduction in caregiver burden) improve AD completion as compared to a no-intervention control group?

Study Design: The project will conduct a 3-group randomized trial in which ADs are provided to hospitalized patients by default in the two treatment groups. When discussing the benefits of AD completion, intervention group A nurses will focus on ADs' potential to promote patients' control over the care they receive. In intervention group B, nurses will focus on the potential for AD completion to reduce caregiver burden. In the control group, patients will receive ADs only if they actively request them (as in standard practice). Specially trained nurses will be responsible for conducting the intervention. Training of RNs will consist of didactic and experiential learning on applying endowment and focusing effect scripts in a consistent manner that are true to the behavioral economic principles. Intervention will occur while in the hospital during which the patient will be presented with one of three options by the RN depending on their random assignment. Patients in both intervention groups will be given an AD by default. Patients who elect to complete an AD can have this completed with RN during the hospitalization or during a separate visit hospital worker who is trained in Advance Care Planning (ACP).

Methodology

Patient Eligibility:

The research RN will complete the "Selection of Patient Form" to determine eligibility for participation in the study (see subjects/sample below). Patients who are determined to be eligible for the study, will be asked if they are willing to participate in the study and asked to sign a consent form .

Intervention:

Patient is assigned into one of the three intervention groups and is provided one of three packets (packet includes script , copy of "Your Health, Your Choice: My Advance Directive", and self-addressed stamped envelope). The RN will provide the designated script regarding advance directives (see "Scripts for Intervention Groups"). Four possible outcomes can occur following this visit: A) patient indicates desire to complete AD while in the hospital; B) patient indicates desire to complete AD with ACP facilitator as separate visit; C) patient elects to complete AD on their own, or D) patient declines to complete AD. A).

Subjects/Sample: Hospitalized patients who reside in the County will be randomized to one of three groups. Eligibility will be determined before discharge. Inclusion criteria are adult patients, 50 years and older, who have a serious, life-limiting illness and require hospitalization (see below). Eligible patients will be identified and selected concurrently from new intakes to Genesys Regional Medical Center.

Inclusion Criteria:

A subject will be eligible for study participation if he/she meets the both 1 & 2 criteria:

1.1 Age 50 years and older 2.0 Subject must have one or more of the following serious life limiting illness that requires hospitalization (as determined from review of medical records and clinical judgment) 2.1. Chronic obstructive pulmonary disease (COPD) or any respiratory (pulmonary) disease that requires home oxygen use (e.g. interstitial lung disease, sleep-disordered breathing), 2.2. End Stage Renal Disease 2.3. Peripheral vascular disease (PVD) 2.4. NYHA Class III or IV Heart Failure (HF) Class III: Marked limitation in activity due to symptoms, even during less-than-ordinary activity, e.g. walking short distances (20-100 m). Comfortable only at rest.

Class IV: Severe limitations. Experiences symptoms even while at rest. Mostly bedbound patients.

2.5. Cancer as a discharge diagnosis (any type) Type: 2.6. Neuromuscular/movement disorders: Myasthenia gravis, ALS, Parkinson's, and Multiple sclerosis

Exclusion Criteria:

A subject will not be eligible for study participation if he/she meets any of the following criteria

3.1. Patient cannot sign legal documents such as consent or AD (Impaired decision-making capacity) 3.2. Previously specified written AD 3.3 Patient previously enrolled in this study.

Data Management and Statistical Analysis:

Sample Size- Calculated on the primary outcome of AD completion rate, the investigators used an estimated baseline completion of 10% for the control group. A two-tailed test for comparing completion rates between a default option and the standard, as well as, comparing the two framing interventions will require a total of 350 participants (125 in each intervention and 100 in the control). This achieves a minimum of 88% power to detect a 15% absolute difference between the groups at alpha of 0.05 and accounts for a 5% attrition rate. The hypothesis that AD completion rates differ by at least 15% between two groups within each arm (default option compared to control; autonomy framing compared to caregiver burden framing) will be analyzed using Chi-square analysis.

Expected Outcomes of the Study:

It is hypothesized that offering patients an AD document (by default), in combination with framing the rationale for AD completion (emphasizing either: A. patient control; or B. reduction in caregiver burden) will improve AD completion as compared to a no-intervention control group.

ELIGIBILITY:
Inclusion Criteria:

* 50 years or older
* One or more of the following:
* Chronic obstructive pulmonary disease
* End stge renal disease
* Peripheral vascular disease
* NYHA class II or V heart failure
* Cancer
* Neuromuscular / movement disorder

Exclusion Criteria:

* Patient referred to palliative care
* Patient has advance directive
* Patient has impaired decision making ability
* Patient previously enrolled in this study

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2014-04; Primary Completion 2017-10 (Actual); Study Completion 2019-10 (Actual)

PRIMARY OUTCOMES:
Advance directive document completion | 1 month
  The number of advance directive documents completed within one month of enrollment.

SECONDARY OUTCOMES:
Advance Directive document completion | 1 year
  The number of advance directive documents completed within one year of enrollment.

OTHER OUTCOMES:
Advance directive communication | 1 year
  The number of patients who discuss advance directives with their family or care giver within one year of enrollment.

CONTACTS AND LOCATIONS:
Overall Officials: Mark E Vogel, PhD, Principal Investigator — Ascension Health; Scott Halpern, MD, PhD, Principal Investigator — University of Pennsylvania; Kimberly R Barber, PhD, Study Director — Genesys Regional Medical Director
Locations (1):
- Genesys Regional Medical Center, Grand Blanc, Michigan, United States